CLINICAL TRIAL: NCT00223925
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Assess the Safety, Tolerability, and Prophylactic Anti-cytomegalovirus Activity of Maribavir in Recipients of Allogeneic Stem Cell Transplants
Brief Title: Maribavir for Prevention of CMV After Stem Cell Transplants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1263-200
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Cytomegalovirus Infection
Keywords: Stem cell transplantation; Allogeneic transplantation
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — maribavir

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Maribavir (100 mg twice daily) (Experimental)
  Interventions: Drug: Maribavir
- Maribavir (400 mg twice daily) (Experimental)
  Interventions: Drug: Maribavir
- Maribavir (400 mg once daily) (Experimental)
  Interventions: Drug: Maribavir

INTERVENTIONS:
Drug: Maribavir
  Arms: Maribavir (100 mg twice daily); Maribavir (400 mg once daily); Maribavir (400 mg twice daily)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Cytomegalovirus (CMV) infections remain a significant problem following various types of transplants that are associated with strong immunosuppressive therapy. Maribavir is a new oral anti-CMV drug with a novel mechanism of action compared to currently available anti-CMV drugs. This study will test the safety and anti-CMV activity of different doses of maribavir when given as CMV prophylaxis following stem cell transplants.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic stem cell transplant recipient
* Recipient CMV seropositive
* Have transplant engraftment
* Able to swallow tablets

Exclusion Criteria:

* CMV organ disease
* HIV infection
* Use of other anti-CMV therapy post-transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2004-10-28 (Actual); Primary Completion 2006-04-05 (Actual); Study Completion 2006-04-05 (Actual)

PRIMARY OUTCOMES:
Clinical safety as measured by the recording of treatment emergent adverse events | 13 weeks

SECONDARY OUTCOMES:
Incidence of CMV disease | 13 weeks
Incidence of CMV infection | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (13):
- United States (13):
  - City of Hope Medical Center, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - Loyola University, Maywood, Illinois
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Wayne State Medical Center, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Medical Center, Durham, North Carolina
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Winston DJ, Young JA, Pullarkat V, Papanicolaou GA, Vij R, Vance E, Alangaden GJ, Chemaly RF, Petersen F, Chao N, Klein J, Sprague K, Villano SA, Boeckh M. Maribavir prophylaxis for prevention of cytomegalovirus infection in allogeneic stem cell transplant recipients: a multicenter, randomized, double-blind, placebo-controlled, dose-ranging study. Blood. 2008 Jun 1;111(11):5403-10. doi: 10.1182/blood-2007-11-121558. Epub 2008 Feb 19. PMID 18285548